CLINICAL TRIAL: NCT07202520
Title: Evaluation of the Benefit of the H'Ability Home Device Used in Supervised Self-rehabilitation at Home on the Autonomy of Post-stroke Patients
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: H'ability (Industry)
Collaborators: Pôle Saint Hélier (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Supportive Care
Other Study IDs: IVR-Home
Record Dates: First submitted 2025-08-08; First posted 2025-10-01 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-09

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Intervention Model Description: After screening visit, patients are randomised between two Arms. Patients in Arm 1 start with experimental phase (H'Ability Home) and after a wash-out period start the control phase (paper). Patients randomised in Arm 2 start with the control phase and after the wash-out period start the experimental phase.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm 1 : IVR + Control (Other): 6 weeks of using H'Ability Home at home (experimental phase) followed by a week of washout and then 6 weeks of using a paper-based exercise guide
  Interventions: Device: IVR : H'Ability Home; Device: Control: paper-based exercise guide
- Arm 2 : Control + IVR (Other): 6 weeks of using a paper-based exercise guide followed by a week of washout and then 6 weeks of using H'Ability Home at home (experimental phase)
  Interventions: Device: IVR : H'Ability Home; Device: Control: paper-based exercise guide

INTERVENTIONS:
Device: IVR : H'Ability Home — H'Ability Home is a Dtx (Digital therapeutics) designed for the neurological rehabilitation of patients who have suffered a stroke, via a wireless virtual reality headset, with a simplified control interface on a tablet or PC
Device: Control: paper-based exercise guide — self-rehabilitation booklet used in current practice in centers
  Other Names: Control

SUMMARY:
The goal of this clinical investigation is to evaluate the benefit of the H'Ability Home device used in supervised self-rehabilitation at home on the autonomy of post-stroke patients.

Participants will perform their self-rehabilitation exercises at home using a virtual reality headset incorporating H'Ability Home software for 6 weeks during the experimental phase. This phase will be compared to a 6-week control phase at home, with self-rehabilitation exercises presented in a paper format.

DETAILED DESCRIPTION:
This is a prospective, multicenter, randomized, controlled, crossover, and repeated-measures clinical study.

Patients with a first stroke, currently undergoing rehabilitation in a center with a planned return home, and with low to reasonable susceptibility to motion sickness will be enrolled.

After inclusion, patients will be randomized to one of two study arms.

* Arm 1: Experimental phase / Washout / Control phase
* Arm 2: Control phase / Washout phase / Experimental phase

During the experimental phase, patients will perform their self-rehabilitation exercises at home using the H'Ability Home device for six weeks.

During the control phase, patients will perform their self-rehabilitation exercises at home using a paper-based exercise guide for six weeks. The two study phases are separated by a one-week washout period during which patients will not perform any self-rehabilitation exercises.

ELIGIBILITY:
Patient Inclusion Criteria:

* Stroke diagnosis: first stroke, with no history of stroke, documented in the medical record
* Currently in rehabilitation (in a center) (full hospitalization or day hospitalization for at least 3 days/week) for another 2 to 4 weeks.
* Planned return home (home self-rehabilitation phase): Patients at the end of their rehabilitation stay and scheduled to return home where the self-rehabilitation phase can take place.
* Ability to use virtual reality: Physical and cognitive ability to interact with virtual reality devices, at the discretion of therapists.
* Adult: Patients aged 18 years or older.
* Informed consent: Voluntary agreement to participate in the study after a full explanation of its terms and conditions.
* Member of a social security scheme or eligible beneficiary
* Distance between home and center included within the usual perimeter of each site.
* Presence of a third-party family caregiver at home who has agreed to ensure the patient's safety during self-rehabilitation sessions with the H'Ability Home device (consent)
* Availability of a Wi-Fi network and internet access at the patient's home
* Presence of an adequate space at home to perform rehabilitation exercises
* Person with low to reasonable sensitivity to motion sickness (MSSQ ≤ 15)

Patient non inclusion Criteria:

* • Visual disorders incompatible with the use of virtual reality (absence of binocular vision, blindness, conjunctivitis, etc.) at the discretion of the investigator. PS: Visual disorders corrected by wearing a vision correction device are not concerned because glasses or contact lenses can be worn when using an IVR headset.

  * Major cognitive impairment: Severe cognitive impairment affecting the patient's ability to understand or follow study instructions, or to operate the device independently, at the investigators' discretion.
  * History of epilepsy: History of epileptic seizures, particularly photosensitive seizures, which may be triggered or aggravated by the use of virtual reality.
  * Medical instability: presence of unstable or uncontrolled medical conditions that could interfere with active participation in rehabilitation.
  * Psychiatric illnesses: active psychiatric disorders (e.g., psychosis, unstabilized bipolar disorder) that could disrupt participation and continuity of rehabilitation, at the investigators' discretion.
  * Wearing implantable medical devices or personal medical devices that could be affected by radio waves (pacemakers, cochlear implants, etc.)
  * Participation in another clinical study: engagement in another clinical study likely to interfere with the study objectives or outcome assessments
  * Planned hospitalization during the home self-rehabilitation period
  * Pregnant, childbirth, or breastfeeding women
  * Persons deprived of their liberty by a judicial (including guardianship, curatorship, and judicial protection) or administrative decision
  * Persons receiving psychiatric care or admitted to a health or social care facility for purposes other than research
  * Persons in an emergency situation unable to express their prior consent

Third-party family caregiver Inclusion Criteria:

* Adult: Person aged 18 years or older
* Informed consent: Voluntary agreement to participate in the study after a full explanation of its terms and conditions.
* Member of a social security scheme or entitled person
* Patient's family caregiver
* Ability to assist the patient in using the device
* Ability to ensure the patient's safety when using the device
* Agreement to assist and ensure the patient's safety when using the device at home
* Agreement to provide feedback on the device by completing self-administered questionnaires (UTAUT) - optional

Third-party family caregiver non-inclusion Criteria:

* Pregnant, childbirth, or breastfeeding women
* Persons deprived of their liberty by a judicial (including guardianship, curatorship, and judicial protection) or administrative decision
* Persons receiving psychiatric care or admitted to a health or social care facility for purposes other than research
* Persons in an emergency situation unable to express their prior consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2025-10-30 (Estimated); Primary Completion 2026-08-08 (Estimated); Study Completion 2026-09-29 (Estimated)

PRIMARY OUTCOMES:
To evaluate the impact of the H'Ability Home device on the level of autonomy of post-stroke patients compared to the exercise booklet. | T0 (screening), T1(Baseline), T2(week 6), T3(week 7), T4 (week 13)
  Level of autonomy by the functional independence measure (FIM) score. From 18 (no autonomy) to 126 (full autonomy).

SECONDARY OUTCOMES:
To evaluate the impact of the H'Ability Home device on the walking speed of post-stroke patients compared to the exercise booklet. | T0 (screening), T1(Baseline), T2(week 6), T3(week 7), T4 (week 13)
  walking speed by the duration of the 10 meters of walking
To evaluate the impact of the H'Ability Home device on the coordination of post-stroke patients compared to the exercise booklet. | T0 (screening), T1(Baseline), T2(week 6), T3(week 7), T4 (week 13)
  coordination by the Quick-DASH score (DASH: Disabilities of the Arm, Shoulder and Hand). scored from 11 (no incapacity) to 100 (full incapacity)
To evaluate the impact of the H'Ability Home device on the quality of life of post-stroke patients compared to the exercise booklet. | T1(Baseline), T2(week 6), T3(week 7), T4 (week 13)
  quality of life by the EuroQoL-5D score. from 1 (no problem) to 5 (extreme problems)
Evaluate the impact of the H'Ability Home device on satisfaction with rehabilitation exercises in post-stroke patients compared to the exercise booklet. | T2(week 6), T4 (week 13)
  satisfaction by the visual digital scale Satisfaction score. From 0 (total insatisfaction) to 10 (total satisfaction)
To evaluate the effect of the H'Ability Home device on the cognitive abilities of post-stroke patients compared to the exercise booklet. | T1(Baseline), T2(week 6), T3(week 7), T4 (week 13)
  cognitive abilities by Mini-Mental State Examination score. From 0 (significant cognitive impairment) to 30 (optimal cognitive abilities)
Evaluate the impact of the H'Ability Home device on the fear of falling in relation to the exercise booklet. | T1(Baseline), T2(week 6), T3(week 7), T4 (week 13)
  fear of falling by the Short-Falls Efficacy Scale-International score scored from 7 (minimal fear) to 28 (maximal fear)
Describe patient compliance with both devices: H'Ability Home and exercise booklet. | T2(week 6), T4 (week 13)
  compliance by number of connections or achievements
Evaluate the acceptability of the H'Ability Home device among patients and caregivers before use (a priori acceptability) and after use (a posteriori acceptability) | T0 (screening), T2(week 6), T4 (week 13)
  acceptability by the score of the Unified Theory of Acceptance and the Use of Technology dimensions. caregiver: from 28 (low acceptance) to 196 (high acceptance). patients: from 31 (low acceptance) to 217 (high acceptance)
Describe the level of mental load of patients with the two devices: H'Ability Home and exercise booklet | T2(week 6), T4 (week 13)
  mental load by NASA Task Load Index score. from 0 (low cognitive load) to 100 (high cognitive load)
Describe the level of motion sickness associated with the use of the H'Ability Home virtual reality device | T2(week 6), T4 (week 13)
  motion sickness by Simulator Sickness Questionnaire score. From 0 (no cinetose) to 48 (severe cinetose)

CONTACTS AND LOCATIONS:
Overall Officials: Emilie LEBLONG, MD, PhD, Principal Investigator — Pôle Saint Hélier
Locations (5):
- France (5):
  - Fondation Hopale - Centre de Jacques Calvé, Berck
  - Hôpital Léon Bérard, Hyères
  - Centre Mutualiste de Rééducation et de Réadaptation Fonctionnelles (CMRRF) de KERPAPE, Ploemeur
  - Pôle Saint Hélier, Rennes
  - Fondation ILDYS - Centre de Perharidy, Roscoff

IPD SHARING:
Plan to Share IPD: No